CLINICAL TRIAL: NCT03902301
Title: The Effect of Lactobacillus Rhamnosus Supplementation on Body Mass, Hyperandrogenism and Insulin Resistance in Overweight and Obese Polycystic Ovary Syndrome Women - Randomized Nutritional Study
Brief Title: Lactobacillus Rhamnosus and PCOS Treatment
Acronym: ProjectPCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Karolina Łagowska, Principal Investigator (dr inż), Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Project PCOS
Record Dates: First submitted 2019-03-11; First posted 2019-04-04 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Insulin Resistance; Polycystic Ovary Syndrome; Hyperandrogenism; Obesity
Keywords: Lactobacillus rhamnosus; Polycystic Ovary Syndrome; insulin resistance; nutrition intervention; probiotic
MeSH Terms: conditions — Insulin Resistance; Polycystic Ovary Syndrome; Hyperandrogenism; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary group (Active Comparator): A diet based on general recommendations for people with insulin resistance for 20 weeks.
  Interventions: Dietary Supplement: Dietary group
- Lactobacillus rhamnosus group (Experimental): Lactobacillus rhamnosus for 20 weeks, (2x 6×10 9 CFU/per capsulex); A diet based on general recommendations for people with insulin resistance.
  Interventions: Dietary Supplement: Lactobacillus group

INTERVENTIONS:
Dietary Supplement: Lactobacillus group — Nutrition intervention focused on the treatment of insulin resistance + Lactobacillus rhamnosus supplementation (6x10 9 of lactobacillus rhamnosus x 2 times a day) (35 people).
  Arms: Lactobacillus rhamnosus group
Dietary Supplement: Dietary group — Nutritional intervention focused on the treatment of insulin resistance (35 subjects).
  Arms: Dietary group

SUMMARY:
The effect of Lactobacillus rhamnosus supplementation on body weight, hyperandrogenism and insulin resistance in overweight and obesity women with Polycystic Ovary Syndrome will be analysed.

ELIGIBILITY:
Inclusion criteria:

* patients diagnosed with PCOS,
* BMI> 28 kg/m2 (overweight or obesity),
* patients not participating in other similar research programs at the same time,
* no previous operations on ovaries such as: laparoscopy, ovarian cautery etc.,
* written agreement to take part in the research.

Exlusion criteria:

* the use of antibiotics or probiotics within 6 months before the start of the experiment,
* the use of pharmacological agents or hormones that may affect the course of the menstrual cycle or metabolic rate within 3 months,
* the use of medicament that may affect on carbohydrate metabolism within 4 weeks,
* failure to comply with dietary recommendations established during the nutritional intervention,
* the use of weight loss supplements during the study,
* clinical diagnosis of digestive disease (for example: irritable bowel syndrome, ulcerative colitis, Crohn's disease, celiac disease),
* pregnancy and breast feeding.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 20 weeks
  Fasting insulin concentration (uU/ml) will be measured before and after 2 hours of 75g glucose drink. Insulin resistance will be measured before and after 20 weeks of the intervention.
Oral glucose test OGTT | 20 weeks
  Fasting glucose concentration (mg/dL) will be measured before and after 2 hours of 75g glucose drink. OGTT will be measured before and after 20 weeks of the intervention. Fating glucose and fasting insulin concentrations will be combined to report HOMA-IR index (homeostatic model assessment of insulin resistance).
Testosterone | 20 weeks
  Testosterone (ng/mL) concentrations will measured at baseline and after 20 weeks of the intervention. Results of testosterone level and SHBG level will be combined to report FAI index (index of free androgen).
DHEA-SO4 | 20 weeks
  DHEA-SO4 (umol/L) concentrations will measured at baseline and after 20 weeks of the intervention. Results of testosterone level and SHBG level will be combined to report FAI index (index of free androgen).
SHBG | 20 weeks
  SHBG (nmol/L) concentrations will measured at baseline and after 20 weeks of the intervention. Results of testosterone level and SHBG level will be combined to report FAI index (index of free androgen).
Free androgen index FAI | 20 weeks
  Results of testosterone level and SHBG level will be combined to report FAI index (index of free androgen).
Body weight | 20 weeks
  Body weight (kg) will be assessment at baseline and after 20 weeks of the intervention.
Body height | Baseline
  Body height (cm) will be assessment at baseline of the intervention.
Body composition | 20 weeks
  Fat mass (%), fat free mass (%) will be assessment at baseline and after 20 weeks of the intervention.
Blood lipid profile: cholesterole | 20 weeks
  Cholesterole (mg/dL) will be measured at baseline and after 20 weeks of the intervention
Blood lipid profile: triglicerydes | 20 weeks
  Triglicerydes (mg/dL) will be measured at baseline and after 20 weeks of the intervention
Blood lipid profile: high density lipoprotein | 20 weeks
  High density lipoprotein HDL (mg/dL) will be measured at baseline and after 20 weeks of the intervention
Blood lipid profile: low density lipoprotein | 20 weeks
  Low density lipoprotein LDL (mg/dL) will be measured at baseline and after 20 weeks of the intervention

SECONDARY OUTCOMES:
Assessment of qualitative and quantitative of the microbiome | 20 weeks
  Qualitative and quantitative determination of the composition of gut microbiota will be assessment at baseline and after 20 weeks of the intervention
Assessment of B-glucuronidase and B-glucosiadase activity | 20 weeks
  B-glucuronidase and B-glucosiadase activity in stoolen sample will be assessment at baseline and after 20 weeks of the intervention
Assessment of short-chain fatty acids | 20 weeks
  Assessment of short-chain fatty acids will be assessment at baseline and after 20 weeks of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland